CLINICAL TRIAL: NCT03540758
Title: Regulation of Endogenous Glucose Production by Central KATP Channels
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Meredith Hawkins (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); American Diabetes Association (Other)
Responsible Party: Sponsor-Investigator, Meredith Hawkins, Principal Investigator, Albert Einstein College of Medicine
Organization: Albert Einstein College of Medicine (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 2018-9039; R01DK069861 (NIH)
Record Dates: First submitted 2018-05-17; First posted 2018-05-30 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Type 2 Diabetes Mellitus; Glucose Metabolism Disorders; Glucose, High Blood
Keywords: type 2 diabetes; diabetes; insulin resistance; diazoxide
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Glucose Metabolism Disorders; Diabetes Mellitus; Insulin Resistance | interventions — Diazoxide; Niacin

STUDY DESIGN:
Who Masked: Participant
Masking Description: The subject will be blinded as to the intervention being received first (Drug or Placebo).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (8):
- Non-diabetic (Diazoxide) (Experimental): Pancreatic clamp study will be done after giving Diazoxide (Proglycem) oral suspension to non-diabetic participants.
  Interventions: Drug: Diazoxide
- Non-diabetic (Placebo) (Placebo Comparator): Pancreatic clamp study will be done after giving a taste-matched placebo for Diazoxide (Proglycem) to non-diabetic participants.
  Interventions: Drug: Placebo
- T2D (Diazoxide) (Experimental): Pancreatic clamp study will be done after giving Diazoxide (Proglycem) oral suspension to type 2 diabetic participants.
  Interventions: Drug: Diazoxide
- T2D (Placebo) (Placebo Comparator): Pancreatic clamp study will be done after giving a taste-matched placebo for Diazoxide (Proglycem) to type 2 diabetic participants.
  Interventions: Drug: Placebo
- T2D (Diazoxide + Nicotinic Acid) (Experimental): Pancreatic clamp study will be done after giving Diazoxide (Proglycem) oral suspension to type 2 diabetic participants after lowering free fatty acids with a nicotinic acid (Niacin) infusion.
  Interventions: Drug: Diazoxide; Drug: Nicotinic acid
- T2D (Nicotinic Acid + placebo for diazoxide) (Experimental): Pancreatic clamp study will be done after lowering free fatty acids with a nicotinic acid (Niacin) infusion in type 2 diabetic participants, and after giving a taste-matched placebo for Diazoxide (Proglycem) to type 2 diabetic participants.
  Interventions: Drug: Nicotinic acid; Drug: Placebo
- Non-diabetic (Diazoxide + Nicotinic Acid) (Experimental): Pancreatic clamp study will be done after giving Diazoxide (Proglycem) oral suspension to non-diabetic participants after lowering free fatty acids with a nicotinic acid (Niacin) infusion
- Experimental: Non-diabetic (Nicotinic Acid + placebo for diazoxide) (Experimental): Pancreatic clamp study will be done after lowering free fatty acids with a nicotinic acid (Niacin) infusion in non-diabetic participants, and after giving a taste-matched placebo for Diazoxide (Proglycem) toon-diabetic participants.
  Interventions: Drug: Nicotinic acid; Drug: Placebo

INTERVENTIONS:
Drug: Diazoxide — Non-diabetic participants will receive diazoxide at a dose of 4-7 mg/kg (based upon weight) before undergoing the pancreatic clamp study.
  T2D participants will have their blood sugar levels normalized, and will then receive diazoxide at a dose of 4-7 mg/kg (based upon weight) before undergoing the pancreatic clamp study.
  Other Names: Proglycem
  Arms: Non-diabetic (Diazoxide); T2D (Diazoxide + Nicotinic Acid); T2D (Diazoxide)
Drug: Nicotinic acid — T2D participants will have their blood sugar levels normalized and will additionally receive nicotinic acid infusion based on weight (0.01 mg/kg/min) to lower free fatty acid levels before undergoing the pancreatic clamp study.
  Other Names: Niacin
  Arms: Experimental: Non-diabetic (Nicotinic Acid + placebo for diazoxide); T2D (Diazoxide + Nicotinic Acid); T2D (Nicotinic Acid + placebo for diazoxide)
Drug: Placebo — Non-diabetic participants will receive placebo and undergo the pancreatic clamp study.
  T2D participants will have their blood sugar levels normalized, and will then receive a taste-matched placebo for diazoxide before undergoing the pancreatic clamp study.
  Other Names: Control
  Arms: Experimental: Non-diabetic (Nicotinic Acid + placebo for diazoxide); Non-diabetic (Placebo); T2D (Nicotinic Acid + placebo for diazoxide); T2D (Placebo)

SUMMARY:
Type 2 diabetes (T2D) affects the ability of the body to process glucose (sugar). Under fasting conditions, the liver is able to make sugar to maintain glucose levels in an important process called endogenous glucose production (EGP). Previous studies suggest that the central nervous system (CNS), including the brain, helps to regulate levels of glucose in the body by communicating with the liver. This process can be impaired in people with type 2 diabetes, and can contribute to the high level of glucose seen in these individuals.

The purpose of this study is to understand how activating control centers of the brain with a medication called diazoxide can affect how much glucose (sugar) is made by the liver. This is particularly important for people with diabetes who have very high production of glucose, which in turn can lead to diabetes complications.

DETAILED DESCRIPTION:
In this study, the investigators will study healthy participants and participants with type 2 diabetes through a procedure called a "pancreatic clamp" study. During the clamp procedure, glucose (a sugar) and insulin (a hormone produced in the pancreas that regulates the amount of glucose in the blood) are infused with an intravenous catheter, and blood samples are collected periodically throughout the procedure to measure blood sugar levels and the levels of several hormones that are found in the body and are related to glucose metabolism. Endogenous glucose production (a measure of the body's production of sugar) will be measured in patients given diazoxide (a medication that activates potassium channels in the brain that may affect glucose production in the liver through brain-liver signaling), compared with when a placebo is given. This study will also investigate whether lowering free fatty acid levels which may help improve the body's ability to regulate glucose levels.

Aim 1: non-diabetic participants will be studied after receiving diazoxide or placebo in a randomized, single-blinded fashion to determine whether extra-pancreatic KATP channels regulate hepatic glucose fluxes in non-diabetic humans.

For Aim 1, 15 healthy, non-diabetic individuals will be studied under the following experimental conditions, in random order and in double blinded fashion:

1. normoglycemic 'pancreatic clamp' studies with administration of placebo
2. normoglycemic 'pancreatic clamp' studies with administration of diazoxide

   Aim 2: participants with type 2 diabetes will be studied after receiving diazoxide or placebo in a randomized, single-blinded fashion to establish whether central regulation of glucose production is impaired in patients with T2D

   For Aim 2, the study population will consist of 15 subjects with moderate-to-poorly controlled Type 2 Diabetes Mellitus (HbA1c 8-12%). In these studies, the effects of diazoxide on EGP under the following 2 experimental conditions will be examined, on separate occasions at least 3 weeks apart, in random order and in double blinded fashion:
3. normoglycemic 'pancreatic clamp' studies with administration of placebo
4. normoglycemic 'pancreatic clamp' studies with administration of diazoxide

Aim 3: participants with type 2 diabetes will be studied after receiving diazoxide or placebo in a randomized, single-blinded fashion after lowering their free fatty acid (FFA) levels to determine whether central regulation of glucose fluxes can be restored upon lowering FFA levels in T2D.

Chronic, moderate increases in FFA levels characteristic of T2D can increase EGP through multiple effects on hepatic glucose fluxes, which may overwhelm the effects of activating central KATP channels. 15 nondiabetic and 15 T2D subjects will be studied under baseline conditions and following nicotinic acid administration, under the following experimental conditions. EGP will be assessed in each subject on separate occasions, at least 3 weeks apart. Placebo and diazoxide will be administered in random order and in double blinded fashion. Heart rate variability may be assessed as a measure of vagal nerve activation:

1. normoglycemic (90 mg/dl) pancreatic clamp studies will be performed following nicotinic acid administration, and placebo
2. normoglycemic (90 mg/dl) pancreatic clamp studies will be performed following nicotinic acid administration, and diazoxide

ELIGIBILITY:
Inclusion Criteria:

For healthy participants:

* Age: 21-70 years old
* Body Mass Index (BMI) under 35
* Negative drug screen
* Normal Hemoglobin A1c (HbA1c) and fasting glucose
* No family history of diabetes among first degree relatives (e.g., mother, father)

For T2D participants:

* Age: 21-70 years old
* BMI under 35
* Stable and moderate-to-poor glycemic control (HbA1c: 8.0-12.0%)
* Negative drug screen
* Not suffering from a previously diagnosed proliferative retinopathy, significant diabetic renal disease or severe neuropathy (including cardiovascular and gastrointestinal autonomic dysfunction).

Exclusion Criteria:

* Age: Under 21 or over 70 years ol
* BMI: >35 for Type 2 Diabetes (T2D) and Non-Diabetic (ND) subjects
* Blood pressure >150/90 or <90/60 on more than one occasion
* Severe polydipsia and polyuria (in subjects with T2D). Since polydipsia and polyuria are common symptoms of T2D, the distinction "severe" denotes that the subject indicates a worsening in the symptoms and/or an experience of discomfort related to the symptoms at the time of screening and/or at the time of withdrawal from the medications
* Urine microalbumin: >300 mg/g of creatinine (in subjects with T2D)
* Uncontrolled hyperlipidemia defined as Triglycerides (TG) > 400 mg/dL and/or Total Cholesterol >300 mg/dL
* Clinically significant liver dysfunction including thrombocytopenia (platelets <100,000/uL), anemia (as below), hypoalbuminemia (<3.5 g/dL), coagulopathy (INR > 1.5), and/or liver enzymes more than 3 times the upper limit of normal
* Clinically significant kidney dysfunction, Glomerular Filtration Rate (GFR): <60 mg/dL
* Clinically significant anemia Prospective subjects with hemoglobin below the lower limit of 12 g/dl for for men and 11 g/dL for women will be assessed with history and physical exam to rule out clinically significant anemia, defined as an individual with symptoms (e.g., fatigue, weakness, shortness of breath, palpitations), signs (pallor, brittle nails etc.), or currently under treatment for anemia. In the absence of a documented hemoglobin decrease or iron deficiency, subjects will not be excluded
* Clinically significant leukocytosis or leukopenia
* Clinically significant thrombocytopenia or thrombocytosis
* Coagulopathy
* Urine drug screen positive for any of the following: amphetamines, barbiturates, benzodiazepines, cocaine, methadone, opiates, oxycodone, phencyclidine (PCP). Amphetamines, oxycodone, opiates, methadone, and benzodiazepines have been shown to affect glucose metabolism (increased glycemia, increased fasting insulin levels, delayed insulin response to food ingestion, insulin deficiency). As the drug test available in the Clinical Research Center (CRC) is a 7-drug panel, we cannot specifically choose which drugs are screened for. Additionally, in the interest of selecting patients on the basis of their reliability and dependability, we would like to exclude participants using illicit drugs. Occasional use of cannabis (once or twice per week) is not an exclusion factor. If the test is read as "indeterminate" it will be repeated at the bedside and an additional sample will be sent to the lab. Decision to enroll subject that day prior to results from lab being available will be decided on a case-by-case basis, i.e., when all previous drug testing had been negative and clinical suspicion is very low
* Urinalysis: Clinically significant abnormalities
* Clinically significant electrolyte abnormalities
* Smoking >10 cigarettes/day
* Alcohol: Men >14 drinks/week or >4 drinks/day, Women >7 drinks/week or >3 drinks/day
* History of chronic liver disease, active hepatitis infection, HIV/AIDS, chronic kidney disease (stage 3 or greater), active cancer, cardiovascular disease or other heart disease, systemic rheumatologic conditions, seizures, bleeding disorders, muscle disease
* Surgeries that involve removal of endocrine glands except for thyroidectomy (if euthyroid on thyroid hormone replacement - if such history free thyroxine (fT4) and Thyroid Stimulating Hormone (TSH) will be checked)
* Pregnant women
* Subject enrolled in another study less than one month prior to the anticipated start date of the proposed study, besides those done by our group
* Family history of premature cardiac death
* Allergies to medication administered during study
* Uncontrolled psychiatric disorders
* Any condition which in the opinion of the PI makes the subject ill suited for participation in the study

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Change in Endogenous glucose production (EGP) rate | 7 hour infusions, 4 days in total, separated at least 1 month apart, up to 1 year duration
  Rates of EGP (a measure of the body's production of sugar) will be measured using analysis of blood samples taken throughout the pancreatic clamp procedure under various treatment conditions (e.g., placebo, diazoxide, nicotinic acid, nicotinic acid/diazoxide), by monitoring changes in the level of a non-radioactive, naturally occurring form of glucose (sugar). Measurement of blood glucose concentrations will either be performed with a Precision Xceed Pro glucometer (for overnight admissions in subjects with T2D) or an Analox glucose analyzer in the study room. Increased EGP is the major cause of fasting hyperglycemia. EGP will be determined by subtracting the rates of glucose infusion from the tracer-derived Rates of glucose appearance (Ra). Rates of change in EGP will be reported in concentration/time and summarized by study arm using basic descriptive statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Meredith Hawkins, M.D., M.S., Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Albert Einstein College of Medicine, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No